CLINICAL TRIAL: NCT04232332
Title: The Phase I Study of Recombinant Human Nerve Growth Factor Injection in Healthy Chinese Volunteers on Safety, Tolerability and Pharmacokinetics: Randomized, Double-blind, Placebo-controlled, Single / Multiple Dose
Brief Title: The Phase I Study of Recombinant Human Nerve Growth Factor Injection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: PR-JSZX-2019015F
Record Dates: First submitted 2020-01-12; First posted 2020-01-18 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Injury of Optic Nerve
MeSH Terms: conditions — Optic Nerve Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- 3.75μg (pre test) (Experimental): Single dose
  Interventions: Drug: Recombinant human nerve growth factor injection,experimental
- 7.5μg (Experimental): Single dose
  Interventions: Drug: Recombinant human nerve growth factor injection,experimental
- 15μg single dose (Placebo Comparator): Intramuscular injection once
  Interventions: Drug: Recombinant human nerve growth factor injection,single dose
- 30μg single dose (Placebo Comparator): Intramuscular injection once
  Interventions: Drug: Recombinant human nerve growth factor injection,single dose
- 45μg single dose (Placebo Comparator): Intramuscular injection once
  Interventions: Drug: Recombinant human nerve growth factor injection,single dose
- 60μg single dose (Placebo Comparator): Intramuscular injection
  Interventions: Drug: Recombinant human nerve growth factor injection,single dose
- 75μg single dose (Placebo Comparator): Intramuscular injection
  Interventions: Drug: Recombinant human nerve growth factor injection,single dose
- 90μg single dose (Placebo Comparator): Intramuscular injection once
  Interventions: Drug: Recombinant human nerve growth factor injection,single dose
- 30μg multiple dose (Placebo Comparator): The dosage will be adjusted according to the actual situation of the trial
  Interventions: Drug: Recombinant human nerve growth factor injection,multiple dose
- 45μg multiple dose (Placebo Comparator): The dosage will be adjusted according to the actual situation of the trial
  Interventions: Drug: Recombinant human nerve growth factor injection,multiple dose

INTERVENTIONS:
Drug: Recombinant human nerve growth factor injection,experimental — Intramuscular injection once on the first day according to dose requirements
  Other Names: Experimental
  Arms: 3.75μg (pre test); 7.5μg
Drug: Recombinant human nerve growth factor injection,single dose — Intramuscular injection once on the first day according to dose requirements
  Other Names: Placebo
  Arms: 15μg single dose; 30μg single dose; 45μg single dose; 60μg single dose; 75μg single dose; 90μg single dose
Drug: Recombinant human nerve growth factor injection,multiple dose — Intramuscular injection once daily for 7 days according to dose requirements
  Other Names: Placebo
  Arms: 30μg multiple dose; 45μg multiple dose

SUMMARY:
A randomized, double-blind, placebo-controlled, single/multiple dose study of recombinant human nerve growth factor injection in healthy Chinese volunteers on safety, tolerability and pharmacokinetics

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, single / multiple dose trial. recombinant human nerve growth factor injection in healthy Chinese volunteers on safety, and pharmacokinetics.The volunteers will be given the drug by intramuscular injection. The main purpose of this trial is to investigate the safety, tolerability , pharmacokinetics and immunogenicity of Chinese healthy volunteers after intramuscular injection of recombinant human nerve growth factor injection, to provide a safe dose range for subsequent clinical trials, as well as a safe and reasonable drug delivery program.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-45 years old, including boundary value;
2. The body weight meets the standard, the body weight of male volunteers is not less than 50kg, the body weight of female volunteers is not less than 45kg, the body mass index is in the range of 19-24kg / m2, the body mass index = body weight (kg) / height (M2);
3. volunteers participated in the study voluntarily and signed informed consent.

Exclusion Criteria:

1. Take any prescription or over-the-counter drugs within 2 weeks before screening;
2. Those who have been vaccinated within 3 months before screening;
3. Those who participated in any clinical trial within 3 months before screening;
4. Those who lost blood or donated more than 200 ml blood within 4 weeks before screening or who intend to donate blood during the study or within 4 weeks after the end of the study;
5. Diseases with clinical significance within 2 weeks before screening;
6. Those who had major surgery, trauma or hospitalization within 6 months before screening;
7. There is tattoo or other influence on the injection site to observe the skin condition;
8. Patients with history of central nervous system, mental system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism system, blood system, immune system, endocrine system and skeletal muscle system may endanger the safety of the subjects or affect the research results according to the judgment of the researchers;
9. There is a significant history of allergy in clinic, especially the history of drug allergy, especially the allergy to any component of zx1305 injection;
10. The five items of hepatitis B (hepatitis B surface antigen, hepatitis B surface antibody, hepatitis B e antigen, hepatitis B e antibody, hepatitis B core antibody), hepatitis C antibody, syphilis specific antibody or AIDS joint test have clinical significance;
11. It is suspected that there is alcohol dependence, and the average alcohol intake in the first half year of screening is more than 2 units per day (1 unit = 10ml alcohol, i.e. 1 unit = 200ml beer with 5% alcohol or 25ml spirits with 40% alcohol or 83ml wine with 12% alcohol) or the alcohol test is positive;
12. Those who smoked more than 5 cigarettes per day in the first half year of screening;
13. Those who had a history of drug abuse or had taken drugs within one year before screening, or who were positive in urine test of ketamine, morphine, methamphetamine, dimethyldioxygoamphetamine and tetrahydrocannabinolic acid;
14. Women who are positive in pregnancy, lactation, blood pregnancy or who have not taken effective contraceptive measures in the last month, and men or women who are not willing to take effective non drug contraceptive measures during the whole trial period and who are not willing to take effective contraceptive measures within one year after the end of the trial;
15. The condition of peripheral venous access is poor (difficult to collect blood);
16. There are other reasons that the researchers think should not be selected.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2019-12-26 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Single dose: 28 days / Multiple dose: 34 days
  Record the number of participants with abnormal laboratory values and/or adverse events,calculate frequency and percentage based on correlation with the investigational drug.
Area under curve (AUC) after injection of single dose/multiple dose | Single dose: 24 hours / Multiple doses: 8 days
  To measure the drug concentration in blood samples which collected after injection
Cmax after injection of single dose/multiple dose | Single dose: 24 hours / Multiple doses: 8 days
  To measure the drug concentration in blood samples which collected after injection
Tmax after injection of single dose/multiple dose | Single dose: 24 hours / Multiple doses: 8 days
  To measure the drug concentration in blood samples which collected after injection
T1/2 after injection of single dose/multiple dose | Single dose: 24 hours / Multiple doses: 8 days
  To measure the drug concentration in blood samples which collected after injection

SECONDARY OUTCOMES:
Percentage of Participants With anti-drug antibodies | Single dose: 28 days / Multiple dose: 34 days
  Percentage of participants with treatment-emergent positive anti-drug antibodies was summarized by treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zhao, Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No